CLINICAL TRIAL: NCT05716971
Title: Risk of Retinal Redetachment Under Densiron-68 in Rhegmatogenous Retinal Detachment With Multiple Retinal Breaks: A Retrospective Case Control Study
Brief Title: Redetachment Under Densiron for RD Multiple Breaks
Acronym: Densiron
Status: Completed | Type: Observational
Sponsor: Dar El Oyoun Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Wael Ahmed Ewais, Associate Professor of Ophthalmology Cairo university, Dar El Oyoun Hospital
Other Study IDs: N-123-2022
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Retinal Detachment Multiple Breaks
MeSH Terms: interventions — densiron-68; densiron

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RD: (study case group A): Redetachment under Densiron
  Interventions: Procedure: Densiron-68 (heavy silicone oil) tamponade for retinal detachment
- RA : (control group B): reattachment under Densiron
  Interventions: Procedure: Densiron-68 (heavy silicone oil) tamponade for retinal detachment

INTERVENTIONS:
Procedure: Densiron-68 (heavy silicone oil) tamponade for retinal detachment — pars plana vitrectomy using Densiron-68 at thee end of surgery

SUMMARY:
Densiron is used as a tamponading agent for inferior retinal detachment with inferior retinal breaks However, data about the use of Densiron -68 for RRD with multiple retinal breaks; especially if involving both superior and inferior quadrants; are not sufficient.

DETAILED DESCRIPTION:
Inferior retinal detachment (IRD) (retinal detachment with inferior retinal breaks ± proliferative vitreoretinopathy) poses a challenge to primary pars plana vitrectomy because of the insufficient tamponade effect. Lighter than water tamponading agents - including gas and silicone oil (SO)- provide no contact with inferior retina, which may open up inferior retinal breaks and may develop proliferative vitreoretinopathy (PVR) as well.

Heavier than water tamponading agents are used for IRD with a favorable outcome. They include: fluorosilicone oil (FSO) 1 2, perfluorocarbon liquids 3 4 , semifluorinated alkanes namely perfluorhexyloctane (F6H8) 5, and fluorinated alkanes which include: HeavySil 6, Oxane HD 7 8 9 10, HWS 46-3000 11, and Densiron-68. 12-22

Densiron-68 (Fluoron, Neu Ulm, Germany) consists of a mixture of polydimethylsiloxane 5000 (PDMS) (69.5%) and perfluorhexyloctane (H6F8) (30.5%). It has a viscosity of 1387 mPas, specific gravity of 1.06 g/cm3, and interfacial tension of 35 mN/m. it has been successfully employed for IRD with a favorable outcome. 15,17,19,20,22,16,12-14,23,18 The final retinal reattachment rate reached up to 95%. 15 There are several reports about the use of Densiron-68 for IRD associated with PVR which reveal a favorable secondary reattachment rate; ranging between 70% and 95%. 17,21,24,25

However, data about the use of Densiron -68 for RRD with multiple retinal breaks; especially if involving both superior and inferior quadrants; are not sufficient.

ELIGIBILITY:
Inclusion Criteria:

* - RRD with multiple retinal breaks (MRBs), using Densiron-68 tamponade.
* Age= 16 and older

Exclusion Criteria:

* - RRD using conventional silicone oil (SO) or Gas tamponade.
* RRD with single RBs
* Age < 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of records of cases of "Rhegmatogenous Retinal Detachment (RRD)with multiple Retinal breaks (MRBs) ", for whom pars plana vitrectomy using Densiron-68 as a tamponading agent had been performed, in the period from March 2014 till November 2019
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Number of retinal breaks | 1 month
  ( 2, 3, 4, or more)
Distribution of retinal breaks | 1 month
  superior and inferior / inferior only

SECONDARY OUTCOMES:
RD Quadrants | 1 month
  (1-4)
PVR | 1 month
  (yes / No)
- Hypotony (IOP < 6 mmHg) (yes/ no) - Hypotony (IOP < 6 mmHg) (yes/ no) - Hypotony (IOP < 6 mmHg) (yes/ no) Hypotony (IOP < 6 mmHg | 1 month
  yes / no

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy faculty of medicine, Cairo, Egypt